CLINICAL TRIAL: NCT05095649
Title: Phase II Trial of Donor Regulatory T-cells for Steroid-Refractory Chronic Graft-versus-Host-Disease in Patients Who do Not Obtain Complete Remission With Ruxolitinib
Brief Title: Donor Regulatory T-cells for cGVHD in Patients Who do Not Obtain Complete Remission With Ruxolitinib
Acronym: Treg4GVHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Treg4GVHD
Record Dates: First submitted 2021-05-26; First posted 2021-10-27 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Graft vs Host Disease
Keywords: Ruxolitinib; T cells

STUDY DESIGN:
Intervention Model Description: The doses of Treg-enriched cells will be 2x10^6 cells/kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regulatory T-cell enriched infusion (Experimental): The doses of Regulatory T-cell enriched infusion will be 2x10^6 cells/kg
  Interventions: Biological: Regulatory T-cell enriched infusion

INTERVENTIONS:
Biological: Regulatory T-cell enriched infusion — Enrichment of cluster of differentiation 25hi regulatory T cells from cluster of differentiation antigen 8 and/or cluster of differentiation antigen19 pre-depleted leukapheresis products.

SUMMARY:
Phase II clinical trial to assess the efficacy of donor regulatory enriched T cells in steroid-refractory chronic graft versus host disease patients who did not obtain complete remission under treatment with ruxolitinib

DETAILED DESCRIPTION:
A number of 15 patients will be included to assess the efficacy of donor regulatory enriched T cells in steroid-refractory chronic graft versus host disease patients who did not obtain complete remission after 12 weeks of treatment with ruxolitinib.

The doses of Treg-enriched cells will be 2x10^6 cells/kg.

Survival at 1 year after Treg infusion will be represented based on the clinical data with Kaplan Meier curves.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of allogeneic hematopoietic stem cell transplantation
* Participants must have steroid-refractory cGVHD and had obtained any response other than progression after at least 12 weeks of treatment with ruxolitinib. Steroid-refractory cGVHD is defined as having persistent signs and symptoms of cGVHD despite the use of prednisone at ≥ 0.25 mg/kg/day (or 0.5 mg/kg every other day) for at least 4 weeks (or equivalent dosing of alternate glucocorticoids) without complete resolution of signs and symptoms.
* Stable dose of glucocorticoids for 4 weeks prior to enrollment.
* No addition or subtraction of other immunosuppressive medications (e.g., calcineurin-inhibitors, sirolimus, mycophenolate-mofetil) for 4 weeks prior to enrollment. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range of that drug.
* No age limit. In the case of children participating in the study, the informed consent will be signed by a parents or legal guardians.
* Eastern Cooperative Oncology Group scale performance status 0-2
* Participants must have adequate organ function
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Ongoing prednisone requirement >1 mg/kg/day (or equivalent).
* Concurrent use of calcineurin-inhibitor plus sirolimus (either agent alone is acceptable).
* History of active thrombotic microangiopathy, hemolytic-uremic syndrome or thrombotic thrombocytopenic purpura in the last 6 months.
* New immunosuppressive medication in the 4 weeks prior to enrollment.
* Extra-corporeal Photopheresis or rituximab therapy in the 4 weeks prior to enrollment.
* Post-transplant exposure to T-cell or interleukin-2 targeted medication within 100 days prior to enrollment.
* Donor lymphocyte infusion within 100 days prior to enrollment.
* Active malignant relapse.
* Active uncontrolled infection.
* Organ transplant (allograft) recipient.
* HIV-positive individuals on combination antiretroviral therapy are ineligible.
* Individuals with active uncontrolled hepatitis B or C are ineligible as they are at high risk of lethal treatment-related hepatotoxicity after hematopoietic stem cell transplant.
* Other investigational drugs within 4 weeks prior to enrollment, unless cleared by the Principal Investigator.
* Pregnant women are excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with overall response rate. | 6 months post-infusion
  Obtain ≥65% the overall response rate at 6 months after infusion
Number of Participants with overall response rate. | 1 year post-infusion
  Obtain ≥75% the overall response rate at 1 year after infusion
Survival | 1 year after Regulatory T-cell enriched infusion
  Number of patients who survive after Regulatory T-cell enriched infusion

SECONDARY OUTCOMES:
Disease evaluation through Symptoms of the disease | Screening, weeks 1, 2, 4, 6, 12 and months 6, 9 and 12 months after infusion
  Symptoms of the disease through chronic graft-versus-host disease activity assessment (clinician) according to NIH consensus- form A
Disease evaluation through measurement of quality of life | Screening, weeks 1, 2, 4, 6, 12 and months 6, 9 and 12 months after infusion
  Measurement of quality of life through Functional Assessment of Cancer Therapy - Bone Marrow Transplantation
Disease evaluation through Symptoms of the disease | Screening, weeks 1, 2, 4, 6, 12 and months 6, 9 and 12 months after infusion
  Symptoms of the disease through chronic graft-versus-host disease symptom scoring scale
Immunosuppressive requirements. | Screening, month1, months 3, 6, and 12 after infusion
  Evaluation of needs of additional permitted immunosuppressive treatment administered as concomitant medication
Free survival | 1 year after infusion.
  To evaluate failure free survival (change of immunosuppression, mortality or relapse)
Immunologic monitoring and in vivo Treg tracking through immune globulins | 1 year after infusion and after infusion
  Quantitative immune globulins
Immunologic monitoring and in vivo Treg tracking through plasma | 1 year after infusion and after infusion
  Plasma banking
Immunologic monitoring and in vivo Treg tracking through mononuclear cells | 1 year after infusion and after infusion
  Storage of additional mononuclear cells
Immunologic monitoring and in vivo Treg tracking through lymphocyte | 1 year after infusion and after infusion
  Detailed immunological evaluation of lymphocyte
Immunologic monitoring and in vivo Treg tracking through Natural Killer cell subsets | 1 year after infusion and after infusion
  Quantitative Natural Killer cell subsets
Purity of Treg-enriched cell infusion | Before 24 hours to infusion up infusion day
  Percentage of cells viability, negative gram stain/endotoxin, percentage of cluster of differentiation 4+ cluster of differentiation 25+ cells and cluster of differentiation 4+cluster of differentiation25+cluster of differentiation127- Treg in order to consider for the infusion.
Toxicity monitoring of Treg-enriched cells | Weeks 1, 2, 4, 6, 12 and months 6, 9 and 12 after infusion
  Number of grade 3 or higher Adverse Events and all Serious Adverse Events according to the Version 5.0 of the NCI Common Terminology Criteria for Adverse Events.
Life-threatening infections | Weeks 1, 2, 4, 6, 12 and months 6, 9 and 12 after infusion
  Number of infections
Predictors of clinical response | 1 year after infusion
  Quantify predictors of clinical response among patients receiving ruxolitinib

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Pérez-Simón, M.D. Ph.D, Principal Investigator — Department of Hematology, Hospital Universitario Virgen del Rocío, Sevilla.
Locations (1):
- José Antonio Pérez Simón, Seville, Spain

IPD SHARING:
Plan to Share IPD: No